CLINICAL TRIAL: NCT04258475
Title: The Influence of Concurrent Oral Calcium Carbonate Supplementation on Steady State Pharmacokinetics of Oral Raltegravir.
Acronym: RCPK
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20190750-01H
Record Dates: First submitted 2020-02-03; First posted 2020-02-06 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Calcium Supplementation in HIV Patients Using Raltegravir
Keywords: Raltegravir; Calcium; PK
MeSH Terms: interventions — Tablets; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Raltegravir-Calcium PK measure (Experimental): Period 1: Raltegravir 1200 mg alone; Period 2: Calcium carbonate antacid 500 mg and 1200 mg of raltegravir given concomitantly; Period 3: two tablets of calcium carbonate antacid 500 mg and 1200 mg of raltegravir given concomitantly.
  Patients will have a total of 8 visits during the study. Day 1 visit: Raltegravir 1200 mg oral daily until day 7. Day 7 visit: Timed serial phlebotomy before dosing t(0) and 0.5, 1, 1.5, 2, 3, 4, 6 hours after observed dosing.
  Day 8 visit: 24 h PK sampling followed by Raltegravir 1200 mg + Calcium carbonate 500 mg oral daily until day 14.
  Day 14 visit: Timed serial phlebotomy before dosing t(0) and 0.5, 1, 1.5, 2, 3, 4, 6 hours after observed dosing.
  Day 15 visit: 24 h PK Sampling followed by Raltegravir 1200 mg + Calcium carbonate 1000 mg oral daily until day 21.
  Day 21 visit: Timed serial phlebotomy before dosing t(0) and 0.5, 1, 1.5, 2, 3, 4, 6 hours after observed dosing.
  Day 22 visit: 24 h PK Sampling. Day 51 visit: Final safety visit.
  Interventions: Drug: Raltegravir standard dosage of 1200 mg (two 600 mg tablets) orally once daily.; Drug: Calcium carbonate antacid tablet

INTERVENTIONS:
Drug: Raltegravir standard dosage of 1200 mg (two 600 mg tablets) orally once daily. — Raltegravir will be dosed in a fasted state in all periods. Participants will take Raltegravir along with other ART medication.
  Other Names: RAL; Isentress®
Drug: Calcium carbonate antacid tablet — PK analysis of different doses of calcium carbonate antacid in patients undergoing ART treatment for HIV using Raltegravir.
  Other Names: TUMS® Ultra Strength (US) 500 mg

SUMMARY:
The purpose of this study is to measure change in raltegravir serum pharmacokinetics in steady state, when co-administered with calcium carbonate formulated as antacid.

DETAILED DESCRIPTION:
Raltegravir (Isentress®) is a familiar, well-tolerated oral HIV integrase inhibitor drug. This class of HIV integrase inhibitor drug is a preferred component of combination anti-retroviral therapy (ART). Calcium supplementation is sometimes recommended for persons with HIV due to risk of bone mineral density loss associated with aging and with other medications, including ART. Due to the chemical structure of raltegravir, which contains two metal-binding motifs, drug-drug interactions can occur when co-administered with divalent metal cations. This interaction can lead to the chelation of the drug and a reduction in drug absorption. Previous work reported a notable decrease in oral absorption when raltegravir was administered concomitantly with a 3,000 mg dose of calcium carbonate antacid. Given that current standard daily calcium typically consists of 1000 mg elemental calcium, the proposed study will investigate the impact of a lower dose (500 and 1,000 mg) of calcium carbonate antacid as TUMS® on the pharmacokinetics of a 1200 mg raltegravir once daily dose.

The patient population will consist of volunteers who are taking ART with good virological and immunological effect, and are willing and able to separate once-daily ART dosing from study medications of raltegravir and calcium, by taking other medications in the evening and study medications in the morning, at least 8 hours apart.

This study consists of three periods: Period 1) Each study participant will take two oral raltegravir 600 mg tablets with breakfast once daily alone for 7 days and have serial PK measures of drug levels from serial phlebotomies over 6 hours and at 24-hour follow-up prior to next daily dosage. Period 2) Starting day 8, participants will take the two raltegravir 600 mg tablets orally concurrent with 500 mg calcium carbonate antacid daily, and similarly have PK as on days 7/8 prior, on days 14/15. Period 3) Starting on day 15, participants will take the two tablets of raltegravir 600 mg concurrent with 1,000 mg calcium carbonate antacid daily and have PK as before on days 21/22.

The primary objective of this study is to measure and compare the minimum serum concentration of raltegravir at 24 hours (C24h) from daily dosing in the steady state, after raltegravir administration alone, and with calcium carbonate 500 mg and 1000 mg. A secondary objective is to determine full serum pharmacokinetic measures, for area-under-the-time-concentration curve from 0 to 24 (AUC0-24h) hours, time to and maximum concentration (Tmax and Cmax) and elimination half-life (t1/2).

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be a healthy HIV infected male or female.
2. Patient must be between the ages of 18 and 65.
3. Patient must be undergoing stable effective ART and must be compatible with once a-day study raltegravir or be separable from study calcium co-administration by at least 8 hours in a twice-a-day dosing schedule.
4. Patient must have a viral load < 50 copies/mL within 3 months of study Day 1.
5. Patient must be medically stable at time of study, with no evidence of acute illness as per physician assessment.
6. Patient must be able to read, understand and sign a written informed consent prior to initiation of the study.
7. Patients must be willing to stop using any herbal or natural health products for 2 weeks prior to Day 1 and during the study.

Exclusion Criteria:

1. Patient on any medications that can alter the drug absorption of study medications other than oral contraception and stable effective ART. This includes no micronutrient mineral and trace element supplementation (except calcium).
2. Patient donated blood with the 30 days prior to study start.
3. Persons with prior gastric or enteric surgery, acute medical illness, or anticipated use of other medications, supplements or treatments.
4. Patient has a BMI > 30
5. Patient is unable to understand, consent and adhere to study protocol and procedures.
6. Women who are pregnant, breast-feeding, and not willing to practice contraception during the study period plus one month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-12-09 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Steady-state serum pharmacokinetics analysis of raltegravir in patients undergoing ART treatment (with raltegravir) and concurrent calcium supplementation. | 22 days
  Determine the minimum (C24h) serum concentration in the steady state of raltegravir 24 hours after dosing of raltegravir 1200 mg alone and when administered concomitantly with calcium carbonate 500 mg or 1000 mg.

SECONDARY OUTCOMES:
Time to peak maximum plasma concentration PK parameter analysis within study duration. | 22 days
  To determine other pharmacokinetic measures including time from observed dosing to maximum plasma concentration, under the same conditions as the primary objectives.
Maximum concentration PK parameter analysis within study duration. | 22 days
  To determine pharmacokinetic measure of maximum concentration under the same conditions as the primary objectives.
Area-under-the-time-concentration curve from 0 to 24 hours PK parameter analysis within study duration. | 22 days
  To determine pharmacokinetic measure of area-under-the-time-concentration curve from 0 to 24 hours under the same conditions as the primary objectives.
Elimination half-life PK parameter analysis within study duration. | 22 days
  To determine pharmacokinetic measure of elimination half-life under the same conditions as the primary objectives.
24-hour concentration (Cmin, Ctrough) of raltegravir PK parameter analysis within study duration within study duration. | 22 days
  To determine pharmacokinetic measure of the 24-hour concentration (Cmin, Ctrough) of raltegravir under the same conditions as the primary objectives.

CONTACTS AND LOCATIONS:
Overall Officials: Bill Cameron, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital General Campus, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Derived] Teixeira Nunes Porto LL, Doyle MA, Zhang G, Tremblay N, Yazji B, Kanji S, Cameron DW. Influence of concurrent oral calcium carbonate supplementation on steady-state pharmacokinetics of once daily oral raltegravir in persons with HIV: a protocol for a prospective open-label non-randomised study in Canada. BMJ Open. 2025 Jul 5;15(7):e094384. doi: 10.1136/bmjopen-2024-094384. PMID 40617620